CLINICAL TRIAL: NCT01535417
Title: A 12 Weeks, Randomized, Double-blind, Multi-centers, Phase III Study to Evaluate the Efficacy and Safety of Shinbaro Capsule Compared With Celebrex Capsule in Patients With Osteoarthritis of Knee
Brief Title: Efficacy and Safety of Shinbaro Capsule
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Green Cross Corporation (Industry)
Responsible Party: Sponsor
Organization: GC Biopharma Corp (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GCSB_P3
Record Dates: First submitted 2012-02-12; First posted 2012-02-17 (Estimated); Last update posted 2012-02-17 (Estimated); Status verified 2012-02

CONDITIONS: Osteoarthritis
Keywords: Osteoarthritis
MeSH Terms: conditions — Osteoarthritis | interventions — shinbaro; Celecoxib

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- GCSB (Experimental)
  Interventions: Drug: Shinbaro Capsule
- Celebrex (Active Comparator)
  Interventions: Drug: Celebrex

INTERVENTIONS:
Drug: Shinbaro Capsule — Herbal drug (Ledebouriellae Radix, Achyranthis Radix, Acanthopanacis Cortex, Cibotii Rhizoma, Glycine Semen, Eucommiae Cortex)
  Arms: GCSB
Drug: Celebrex
  Arms: Celebrex

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of 'Shinbaro Capsule', a new herbal anti-arthritic agent, in patients with osteoarthritis of the knee.

ELIGIBILITY:
Inclusion Criteria:

* age between 35 and 80
* diagnosed with Knee OA based on criteria of ACR and showed ont through I ~ III of Kellgren Stage on radiography
* wuffered constantly with Knee OA for more than 6 months prior to begining the study
* scored more than 30 on total WOMAC scale

Exclusion Criteria:

* had other comorbid orthopedic disease
* had OA of index knee from significant trauma or surgery

Ages: 35 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 198 (Actual)
Dates: Start 2009-05; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
WOMAC change | Baseline, 12 weeks
  WOMAC change

SECONDARY OUTCOMES:
100mm Pain VAS on walking | Baseline, 12 weeks
  change, percent change
PGART | 12 weeks
Adverse Events | 12 weeks